CLINICAL TRIAL: NCT03845621
Title: Effect of Occlusal Accommodation of the Mouthguard on the Degree of Satisfaction of Water Polo Players: A Randomized Crossover Study
Brief Title: Effect of Occlusal Accommodation of the Mouthguard on the Degree of Satisfaction of Water Polo Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Jordi Martinez-Gomis, Associate Professor DDS. PhD, University of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HOUB2018/031
Record Dates: First submitted 2019-01-22; First posted 2019-02-19 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Satisfaction; Quality of Life
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM-OA-OA-CM Sequence (Active Comparator): Use of a conventional custom-made mouthguard (CM) while playing water polo for first and fourth weeks and the occlusal-adjusted custom-made mouthguard (OA) for the second and third weeks.
  Interventions: Device: Conventional Mouthguard; Device: Occlusal-adjusted Mouthguard
- OA-CM-CM-OA Sequence (Active Comparator): Use of an occlusal-adjusted custom-made mouthguard (OA) for the first and fourth weeks and a conventional custom-made mouthguard (CM) while playing water polo for the second and third weeks.
  Interventions: Device: Conventional Mouthguard; Device: Occlusal-adjusted Mouthguard

INTERVENTIONS:
Device: Conventional Mouthguard — Use of a conventional custom-made mouthguard while playing water polo
Device: Occlusal-adjusted Mouthguard — Use of an occlusal-adjusted custom-made mouthguard while playing water polo

SUMMARY:
This study assesses the effect of adjusting the occlusal surface of a custom-made mouthguard on the degree of satisfaction with a mouthguard among water polo players. Twenty-four water polo players will wear a custom-made conventional mouthguard and a custom-made mouthguard with occlusal adjustment, two weeks per mouthguard. They will wear it during training sessions and for competing. The sequence will be randomized to obtain one-half of the participants starting the first week wearing the conventional mouthguard, and the other half wearing the mouthguard with occlusal adjustment. The participants will rate the degree of interference with oral functions or discomfort in reference to speech, breathing, swallowing, gag reflex, fits too tight, fits too loose, aesthetics and athletic performance, in a 10-point scale, considering 0 no discomfort/interference and 10 maximum discomfort/interference. After each session, players also rated the perception of protection, the degree of improvement on athletic performance and the degree of satisfaction in a 10-point scale, considering 0 no protection/satisfaction and 10 maximum protection/satisfaction.

DETAILED DESCRIPTION:
This crossover intervention study aims to assess the effect of adjusting the occlusal surface of a custom-made mouthguard on the degree of satisfaction with a mouthguard among water polo players. Twenty-four water polo players will participate in this randomized crossover trial. Two different custom-made mouth guards will be made for each participant, a conventional one and an occlusal-adjusted mouthguard. Both types of mouthguard will be fabricated using a pressure molding device and 4-mm ethyl vinyl acetate foils. The conventional mouth guards will be made at 2 mm from the full depth of the labial sulcus, covering the second maxillary molar, and with the palatal margin extending 2 mm from the cervical line. To fabricate the occlusal adjusted mouthguard a second 2-mm foil of ethyl vinyl acetate will be formed over the initial 4-mm layer. The maxillary and mandibular casts mounted to an articulator using an inter occlusal record will facilitate the accommodation of the occlusal surface to the antagonistic teeth. The participants will be instructed to wear the mouth guards during training sessions and competitions. The sequence of use will be randomized to obtain one half of the participants beginning the first and the fourth week wearing the conventional mouthguard and the second and the third wearing the occlusal-adjusted mouthguard. The other half will start wearing the first and the fourth week the mouthguard with occlusal-adjusted mouthguard and the second and third week wearing the conventional mouthguard. The participants will evaluate on a 10-point scale for discomfort (gag reflex, fits too tight, fits too loose), interference with functions (speech, breathing, swallowing, aesthetics, and athletic performance), protection, and general satisfaction after each training session or match.

ELIGIBILITY:
Inclusion Criteria:

- Playing in the highest Spanish league of water polo for the season 2018- 2019

Exclusion Criteria:

- Players with dental caries, periodontitis or temporomandibular joint pain

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Degree of satisfaction using a questionnaire | Weeks 1-4
  Participant satisfaction will be assessed by asking the question "How satisfied are you with your mouthguard?" using a 0-10 point scale, considering 0= totally dissatisfied and 10 = totally satisfied. Players rated the mouthguard just after each training session or after each match.

SECONDARY OUTCOMES:
Degree of interference on speech using a questionnaire | Weeks 1-4
  The degree of interference on speech while using the mouthguard will be assessed by asking the question "How much do you think wearing the mouthguard interferes your ability to speech?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of interference on breathing using a questionnaire | Weeks 1-4
  The degree of interference on breathing while using the mouthguard was assessed by asking the question "How much do you think wearing the mouthguard interferes your ability to breath?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of interference on swallowing using a questionnaire | Weeks 1-4
  The degree of interference on swallowing while using the mouthguard will be assessed by asking the question "How much do you think wearing the mouthguard interferes your ability to swallow?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of discomfort regarding the gag reflex using a questionnaire | Weeks 1-4
  The degree of discomfort regarding the gag reflex while using the mouthguard will be assessed by asking the question "How much do you think wearing the mouthguard causes a gag reflex?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of discomfort because the mouthguard fits too tight using a questionnaire | Weeks 1-4
  The degree of discomfort because the mouthguard fits too tight will be assessed by asking the question "How much do you think the mouthguard fits too tight?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of discomfort related to the dislodgement of the mouthguard using a questionnaire | Weeks 1-4
  The degree of discomfort because the mouthguard dislodges will be assessed by asking the question "How much do you think the mouthguard fits too loose?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of interference on aesthetics using a questionnaire | Weeks 1-4
  The degree of interference on aesthetics while using the mouthguard will be assessed by asking the question "How much do you think wearing the mouthguard interferes on aesthetics?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of interference on athletic performance using a questionnaire | Weeks 1-4
  The degree of interference on athletic performance while using the mouthguard will be assessed by asking the question "How much do you think wearing the mouthguard interferes athletic performance?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of protection using a questionnaire | Weeks 1-4
  The degree of protection perceived by the participant will be assessed by asking the question "How much do you feel protected when you are wearing the mouthguard?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of improvement on athletic performance using a questionnaire | Weeks 1-4
  The degree of improvement on athletic performance while using the mouthguard will be assessed by asking the question "How much do you think wearing the mouthguard improves athletic performance?" using a 0-10 point scale (considering 0= anything to 10= very much). Players rated the mouthguard just after each training session or after each match.
Cost-effectiveness analysis by assessing the degree of satisfaction and the cost of the mouthguard | Weeks 0-4
  The time spent in both the laboratory and the clinical setting and the cost of the materials will be considered for the estimation of the cost-effectiveness of the mouthguard. Effectiveness will be considered as the degree of satisfaction with the mouthguard perceived by the participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordi Martinez-Gomis, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Geary JL, Clifford TJ, Kinirons MJ. Occlusal accommodation and mouthguards for prevention of orofacial trauma. Oral Health Prev Dent. 2009;7(1):55-9. PMID 19408816
- [Background] Zamora-Olave C, Willaert E, Montero-Blesa A, Riera-Punet N, Martinez-Gomis J. Risk of orofacial injuries and mouthguard use in water polo players. Dent Traumatol. 2018 Dec;34(6):406-412. doi: 10.1111/edt.12434. Epub 2018 Oct 10. PMID 30156365
- [Background] Gomez-Gimeno A, Zamora-Olave C, Cordobes-Navarro M, Willaert E, Martinez-Gomis J. Satisfaction with shortening the palatal extension of a mouthguard for water polo players: A randomized crossover study. Dent Traumatol. 2019 Apr;35(2):135-141. doi: 10.1111/edt.12455. Epub 2019 Jan 7. PMID 30481393
- [Result] Flores-Figueiras C, Zamora-Olave C, Willaert E, Martinez-Gomis J. Effect of thickness and occlusal accommodation on the degree of satisfaction with mouthguard use among water polo players: A randomized crossover trial. Dent Traumatol. 2020 Dec;36(6):670-679. doi: 10.1111/edt.12583. Epub 2020 Jul 20. PMID 32590885